CLINICAL TRIAL: NCT01268644
Title: Open Label Single Center Pilot Study to Study Teh Effects of Metreleptin Administration in Patients With Type 1 Diabetes Mellitus ( T1DM ).
Brief Title: Effects of Metreleptin in Type 1 Diabetes Mellitus
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor request
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Amylin Pharmaceuticals, LLC. (Industry)
Responsible Party: Principal Investigator, Abhimanyu Garg, Chief, Division Nutrition and Metabolic Diseases, Professor Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FBA937; CTRC # 953 (Other Grant/Funding Number: JDRF and Amylin)
Record Dates: First submitted 2010-12-29; First posted 2010-12-31 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-07

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Leptin; metreleptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- active open label Leptin (Experimental): Active open label Leptin for type 1 Diabetes
  Interventions: Drug: Leptin

INTERVENTIONS:
Drug: Leptin — weight based sub-cutaneous injection twice daily of Leptin
  Other Names: Metreleptin

SUMMARY:
This study will add leptin therapy to the current insulin therapy of Type 1 Diabetics with the aim of lowering the total insulin requirements and suppressing the steep fluctuations typically associated with Type 1 Diabetes.

DETAILED DESCRIPTION:
The adipocyte hormone, leptin, has been shown to restore the health and glucoregulation of near-death, insulin deficient diabetic rodents. This makes leptin the only hormone, since the discovery of insulin in 1922, with this capability. Leptin normalizes the hyperglucagonemia of diabetes and reduces lipogenesis and cholesterologenenesis. Treatment of diabetic rodents with a combination of leptin and insulin, leads to a stable pattern of glucose control with reduced insulin requirements, as opposed to the high glucose variability that characterizes the treatment of type 1 diabetes with supraphysiologic doses of insulin alone. As such, we will initiate a pilot clinical trial to test combination leptin and insulin therapy in type 1 diabetes. Fifteen leptin sensitive patients (body mass index <27 kg/m²) with uncontrolled diabetes (HbA1c 7.0 to 10.0 %) will be treated with slightly supraphysiologic doses of recombinant human leptin (Amylin Pharmaceuticals). Subjects will be compared to themselves before and after treatment with leptin. Endpoint variables include HbA1c, change in daily insulin dose, mean and standard deviation of blood glucose from inpatient glucose monitoring and glucose meter download. We will also assess effects of leptin therapy on energy intake as assessed by 3-day food record and body weight and fat by DEXA. Intramyocellular and intrahepatic lipid concentration by 1H-MRS will be assessed before and after 3 months of metreleptin therapy. A satiety analysis will be employed. In addition, plasma hormones and inflammatory biomarkers will be assayed during the course of this study.

ELIGIBILITY:
Inclusion Criteria:

All of the following criteria are to be fulfilled for inclusion of an individual in the study. An eligible individual:

1. Is male or female and is 18 to 50 years of age
2. Has been diagnosed with T1DM for at least 1 year. Diagnosis of T1DM will be based on clinical criteria including: insulin-dependence within 6 months of the onset, history of prior episode of ketoacidosis, previous documentation of positive serum islet cell autoantibodies or low or undetectable serum C-peptide levels.
3. Has an HbA1c 7.0 to 10.0 %, inclusive
4. Currently on insulin pump or on a combination of basal (long-acting insulin preparation) and pre-prandial (short-acting insulin preparation) insulin therapy
5. Is male, or if female of childbearing potential, is non-lactating, and has a negative pregnancy test (human chorionic gonadotropin, beta subunit [βhCG]) result at screening (Visit 1) and Visit 2 regardless of menopausal status (If female and of childbearing potential [including peri menopausal women who have had a menstrual period within one year], must practice and be willing to continue to practice appropriate birth control [defined as a method which results in a low failure rate, i.e., less than 1% per year, when used consistently and correctly, such as implants, injectables, oral contraceptives, some intrauterine contraceptive devices, sexual abstinence, tubal ligation, or a vasectomized partner] during the entire duration of the study.)
6. Has a BMI < 27 kg/m2
7. Has clinical laboratory test values (clinical chemistry, hematology, and urinalysis) judged to be not clinically significant by the investigator at screening (Visit 1)
8. Has a physical examination and electrocardiogram (ECG) with no clinically significant abnormalities as judged by the investigator

Exclusion Criteria:

1. Has a fasting serum triglyceride concentration >400 mg/dL at screening
2. Has hypoglycemia unawareness (Loss of consciousness due to hypoglycemia without preceding symptoms or recent history of blood glucose <50 mg/dl without symptoms)
3. Currently abuses drugs or alcohol, or has a history of abuse that in the investigator's opinion could cause the individual to be noncompliant with study procedures, or has a positive urine screen for drugs of abuse at screening (Visit 1)
4. Has chronic renal insufficiency with serum creatinine > 2 mg/dL
5. Has a history of weight loss (>3%) in the last 3 months
6. Is currently enrolled or plans to enroll in a diet, weight loss, or exercise program
7. Has a sitting blood pressure >160/95 mmHg (either systolic or diastolic) at screening (Visit 1)
8. Has a clinically significant history or presence of any of the following conditions:

   * Active cardio- or cerebrovascular disease
   * Active pulmonary disease
   * Hepatic disease defined as follows:

     * At screening (Visit 1), alanine transaminase (ALT), aspartate transaminase (AST), or alkaline phosphatase > three times the upper limit of normal (elevated Liver Function Test values suggestive of obesity related non-alcoholic fatty liver disease may not be exclusionary)
   * The presence of any other co morbid disorders that, in the opinion of the investigator, would interfere with the subject's compliance of study procedures
   * Clinically significant malignancies within 5 years of screening (Visit 1)
   * Chronic infections (e.g., HIV [human immunodeficiency virus] or tuberculosis)
9. Has received any investigational drug within 30 days or within a period corresponding to five half-lives of that drug, whichever is greater, before screening (Visit 1)
10. Has had major surgery or a blood transfusion within 2 months before screening (Visit 1) or has a hematocrit < 30%
11. Has a known hypersensitivity to any of the components of the study treatment (e.g. has a known hypersensitivity to E. Coli derived proteins
12. Is an immediate family member (spouse, parent, child, or sibling; biological or legally adopted) of personnel directly affiliated with the study at the investigative site, or is personally directly affiliated with the study at the investigative site
13. Is employed by Amylin Pharmaceuticals, Inc., (i.e., an employee, temporary contract worker, or designee responsible for the conduct of the study)
14. Has previously received treatment with recombinant leptin (metreleptin or Fc leptin)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2010-09; Primary Completion 2013-01 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abhimanyu Garg, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Background] Vasandani C, Clark GO, Adams-Huet B, Quittner C, Garg A. Efficacy and Safety of Metreleptin Therapy in Patients With Type 1 Diabetes: A Pilot Study. Diabetes Care. 2017 May;40(5):694-697. doi: 10.2337/dc16-1553. Epub 2017 Feb 21. PMID 28223297

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with T1DM between the 18 and 50 years of age and with a BMI less than 27 kg/m2 and an HbA1c of 7.0-10.0% (53-86 mmol/mol) were eligible for the study.
Groups:
- Leptin Therapy in T1DM Patients: After a 4-week lead-in period, baseline evaluation was conducted at week 0.
Period: Baseline Period (Week 0)
Arm/Group | Leptin Therapy in T1DM Patients
Started | 8
Completed | 8
Not Completed | 0
Period: Phase A (Weeks 0-12) Leptin Therapy
Arm/Group | Leptin Therapy in T1DM Patients
Started | 8
Completed | 8
Not Completed | 0
Period: Phase B (Weeks 12-20) Leptin Therapy
Arm/Group | Leptin Therapy in T1DM Patients
Started | 7 (One subject withdrew after 12 weeks .)
Completed | 7
Not Completed | 0
Period: Phase C (Weeks 20-24) Off Leptin Therapy
Arm/Group | Leptin Therapy in T1DM Patients
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Week 0 (Baseline): After a 4-week lead-in period, baseline evaluation was conducted at week 0.
Arm/Group | Week 0 (Baseline)
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 8
Weight [Mean (Standard Deviation); unit: kg] | 70.7 (5.9)
Leptin [Median (Full Range); unit: ng/mL] | 23 [6 to 34]
Insulin dose [Mean (Standard Deviation); unit: Units/day] | 45.9 (11.5)
HbA1c [Mean (Standard Deviation); unit: % of Hemoglobin] | 7.6 (0.4)

OUTCOME MEASURES:

1. Primary Outcome: HbA1c
Description: Change in Hba1c after 12 weeks on Leptin Therapy compared to Baseline value
Time Frame: Baseline and 12 weeks
Measure: Mean (95% Confidence Interval); unit: % of hemoglobin
Groups:
- Leptin Therapy Week 12: Change in HbA1c after 12 weeks on Leptin Therapy from Baseline.
Arm/Group | Leptin Therapy Week 12
Number analyzed (Participants) | 8
% of hemoglobin | -0.19 [-0.44 to 0.07]
Statistical Analysis 1: Comparison: Leptin Therapy Week 12; Test type: Superiority; p = 0.14, Mixed Models Analysis — P value comparing baseline to week 12

2. Secondary Outcome: Weight
Description: Change in Body Weight after 12 weeks on Leptin Therapy compared to Baseline value
Time Frame: Baseline to 12 weeks
Population: One subject withdrew after 12 weeks.
Measure: Mean (95% Confidence Interval); unit: kg
Groups:
- Leptin Therapy in TIDM Patients: Change in Body Weight after 12 weeks on Leptin Therapy compared to Baseline value
Arm/Group | Leptin Therapy in TIDM Patients
Number analyzed (Participants) | 8
kg | -2.60 [-4.6 to -0.6]
Statistical Analysis 1: Comparison: Leptin Therapy in TIDM Patients; Test type: Superiority; p = 0.01, Mixed Models Analysis — P value comparing week 0 with week 12

3. Secondary Outcome: Insulin Dose
Description: Change in Insulin dose after 12 weeks on Leptin Therapy compared to Baseline value
Time Frame: Baseline to 12 weeks
Population: One subject withdrew after 12 weeks.
Measure: Mean (95% Confidence Interval); unit: units/day
Groups:
- Leptin Therapy in TIDM Patients: Change in Daily insulin dose after 12 weeks on Leptin Therapy compared to insulin dose during the Baseline period
Arm/Group | Leptin Therapy in TIDM Patients
Number analyzed (Participants) | 8
units/day | -5.84 [-10.1 to -1.6]
Statistical Analysis 1: Comparison: Leptin Therapy in TIDM Patients; Test type: Superiority; p = 0.009, Mixed Models Analysis — P value comparing week 0 to week 12

4. Secondary Outcome: Change in HbA1c From Baseline to Week 20 on Leptin Therapy
Description: Change in Hba1c after 20 weeks on Leptin Therapy compared to Baseline value. With ongoing metreleptin therapy, the concomitant basal insulin dose was actively reduced by 50% after week 12.
Time Frame: Baseline to Week 20 (On leptin)
Measure: Mean (95% Confidence Interval); unit: % of Hemoglobin
Groups:
- Week 20 (On Leptin): Change in Hba1c after 20 weeks on Leptin Therapy compared to Baseline value. With ongoing metreleptin therapy, the concomitant basal insulin dose was actively reduced by 50% after week 12.
Arm/Group | Week 20 (On Leptin)
Number analyzed (Participants) | 7
% of Hemoglobin | -0.04 [-0.31 to 0.22]
Statistical Analysis 1: Comparison: Week 20 (On Leptin); Test type: Superiority; p = 0.75, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 24 weeks.
Groups:
- Overall Study: After a 4-week lead-in period, baseline evaluation was conducted at week 0.
Arm/Group | Overall Study
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 1/8
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study (N=8)
Injection site reaction (Infections and infestations) | 1 (1) — One subject withdrew after 12 weeks as a result of injection site reaction.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No